CLINICAL TRIAL: NCT03145259
Title: Evaluation of Bioavailability of Diclofenac Dermal Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HP-00067047
Record Dates: First submitted 2017-05-01; First posted 2017-05-09 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Bioavailability
MeSH Terms: interventions — Transdermal Patch; Solutions

STUDY DESIGN:
Intervention Model Description: The same 12 volunteers received all treatments in three separate study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diclofenac patch (Other): Study Session 1: diclofenac epolamine patches (PK) [51 h study duration]
  Interventions: Drug: Diclofenac Epolamine Patch
- Diclofenac solution (Other): Study Session 2: diclofenac sodium solution (PK) [47 h study duration]
  Interventions: Drug: diclofenac sodium solution
- Diclofenac patch and solution (Other): Study Session 3: diclofenac epolamine patch pieces and diclofenac sodium solution (no PK, for skin tape stripping) [51 h study duration]
  Interventions: Drug: Diclofenac Epolamine Patch; Drug: diclofenac sodium solution

INTERVENTIONS:
Drug: Diclofenac Epolamine Patch — patch
  Other Names: patch
  Arms: Diclofenac patch; Diclofenac patch and solution
Drug: diclofenac sodium solution — solution
  Other Names: solution
  Arms: Diclofenac patch and solution; Diclofenac solution

SUMMARY:
The study will utilize already FDA-approved marketed diclofenac products in healthy adults to generate data for establishing rate of drug delivery comparisons between diclofenac epolamine patches and diclofenac sodium solution in healthy adults and to determine skin concentrations.

DETAILED DESCRIPTION:
The study will utilize already FDA-approved marketed diclofenac products in healthy adults to generate data for establishing rate of drug delivery comparisons between diclofenac epolamine patches and diclofenac sodium solution in healthy adults and to determine skin concentrations. This study supports FDA's continuing effort to identify the most accurate, sensitive, reproducible and efficient methods to evaluate topical dermatological drug products.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant, women who are of any ethnic background between the age of 18 to 45 years old
2. Subjects must be non-smokers (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches or electronic cigarettes) over the previous 2 months and are not currently using tobacco products
3. Provide written informed consent before initiation of any of the study procedures
4. Agree not to participate in another clinical trial/study during the study period or to participate in an investigational drug study for at least 1 month after the last study session
5. Able to adhere to the study protocol and study restrictions
6. Able to participate in all study sessions
7. Has a volar forearm of either at least 24 cm (9.45 inches) in length or of sufficient size that can accommodate the products to be tested in a study area that begins at least 5 cm (1.97 inches) above the wrist and ends a minimum of 0.5 cm (0.197 inches) below the antecubital fossa (i.e., the bend in the arm at the elbow).
8. Subjects have upper arms large enough to allow for placement of two 140 cm2 [21.7 in2] patches (distance from acromion process of the scapula to olecranon process should be a minimum of 35 cm [13.8 inches]; circumference of upper arms should be a minimum of 28 cm [11.02 inches] and 200 cm2 [31 in2] area for application of solution
9. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination and medication history
10. Negative urine drug screening test (cannabinoids, amphetamines, barbiturates, benzodiazepine, cocaine, methadone, opiates, PCP)
11. Have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine transaminase (ALT) and aspartate aminotransferase (AST)
12. Have normal screening laboratories for urine protein and urine glucose
13. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of each study session, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner
14. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 3 months after last study session
15. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute)
16. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-165 mmHg
    * Diastolic blood pressure 60-100 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-20 breaths per minute

Exclusion Criteria:

1. Women who are pregnant, lactating, breast feeding or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of the first day of each study session
2. Smokers (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patch or electronic cigarettes)
3. Participation in any ongoing investigational drug trial/study or clinical drug trial/study
4. History as either reported by the subject or evident to the Medically Accountable Investigator (MAI) of infectious disease or skin infection or of chronic skin disease (e.g., psoriasis, atopic dermatitis)
5. History of diabetes
6. History of significant skin cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and did not involve the investigative sites
7. Body Mass Index (BMI) ≥30 kg/m2
8. History of chronic obstructive pulmonary disease or cor pulmonale, or substantially decreased respiratory reserve, hypoxia, hypercapnia or pre-existing respiratory depression
9. Active positive Hepatitis B, C and/or HIV serologies
10. Positive urine drug screening test
11. Use of chronic prescription medications during the period 0 to 30 days; or over-the-counter medication (e.g. antihistamines, topical corticosteroids) and short term (<30 days) prescription medications during the period 0-3 days before a study session (vitamins, herbal supplements and birth control medications not included)
12. Currently taking daily oral nonsteroidal anti-inflammatory drug [NSAIDs] (aspirin, ibuprofen, naproxen, etc…)
13. Currently taking daily anticoagulants or within the past month prior to entry into the study (warfarin, heparin, rivaroxaban, dabigatran, etc…), ACE-inhibitors, cyclosporine, diuretics, lithium or methotrexate
14. Donation or loss of greater than one pint of blood within 60 days of entry to the study
15. Any prior adverse reaction or hypersensitivity to diclofenac, aspirin, ibuprofen, naproxen or other nonsteroidal anti-inflammatory drug (NSAID), other inactive ingredients in the patch or topical solution or to adhesives or tapes used to cover or tape strip the treatment sites
16. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study
17. Eat or drink anything containing alcohol within 24 hours prior to dose administration
18. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
19. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application site (upper arms/volar forearms), sunburn, raised moles or scars, open sores at application site (upper arms/volar forearms), scar tissue, tattoo, or coloration that would interfere with placement of diclofenac products, skin assessment, or reactions to diclofenac
20. History of asthma or urticaria,, hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function or liver disease
21. History of gastrointestinal bleeding or peptic ulcer disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra L Stinchcomb, PhD, Principal Investigator — University of Maryland Baltimore School of Pharmacy; Hazem E Hassan, PhD, Principal Investigator — University of Maryland Baltimore School of Pharmacy
Locations (1):
- General Clinical Research Center (GCRC) at the University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac: Study Session 1. diclofenac epolamine patch Study Session 2. diclofenac sodium solution Study Session 3. diclofenac epolamine patch pieces and diclofenac sodium solution
Period: Overall Study
Arm/Group | Diclofenac
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diclofenac
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Serum Diclofenac Concentrations
Description: Study Session 1: within 60 min prior to dosing, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 24, 27, 30, 32, 51 h Study Session 2: within 60 min prior to dosing, 1, 2, 3, 4, 5, 6, 7, 23, 26, 29, 31, 47 h Study Session 3: no blood samples obtained
Time Frame: blood samples obtained over 51 hour time period for study session 1 and over 47 hour time period for study session 2; through study completion
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Diclofenac Epolamine Patches: diclofenac epolamine patches
  Diclofenac Epolamine Patch: patch
- Diclofenac Sodium Solution: diclofenac sodium solution
  diclofenac sodium solution: solution
Arm/Group | Diclofenac Epolamine Patches | Diclofenac Sodium Solution
Number analyzed (Participants) | 12 | 12
ng/mL | 5.6 (10.8) | 40.0 (54.3)

ADVERSE EVENTS:
Time Frame: From the beginning of the study (10/04/17) through when the last adverse event resolved (05/15/20) [2 years, 7 months] TDCLO-001 (431 days), TDCLO-003 (156 days), TDCLO-004 (740 days), TDCLO-010 (37 days), TDCLO-011 (162 days), TDCLO-012 (306 days), TDCLO-013 (500 days), TDCLO-016 (76 days), TDCLO-019 (52 days), TDCLO-020 (213 days), TDCLO-024 (79 days), TDCLO-029 (58 days)
Groups:
- Diclofenac Epolamine Patches and Diclofenac Sodium Solution: patch pieces and solution
  Diclofenac Epolamine Patch: patch
  diclofenac sodium solution: solution
Arm/Group | Diclofenac Epolamine Patches | Diclofenac Sodium Solution | Diclofenac Epolamine Patches and Diclofenac Sodium Solution
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Epolamine Patches (N=12) | Diclofenac Sodium Solution (N=12) | Diclofenac Epolamine Patches and Diclofenac Sodium Solution (N=12)
Menstrual flow (General disorders) | 1 (1) | 0 (0) | 0 (0) — light menstrual flow (participant noted different from normal)
decreased blood pressure (Eye disorders) | 5 (5) | 5 (5) | 5 (5)
increased heart rate (General disorders) | 1 (1) | 1 (1) | 0 (0)
raised skin (General disorders) | 0 (0) | 0 (0) | 1 (1)
skin hyperpigmentation (General disorders) | 0 (0) | 1 (1) | 9 (9)
abrasions (General disorders) | 0 (0) | 0 (0) | 1 (1) — from tape strips used for skin tape stripping
scabs (General disorders) | 0 (0) | 0 (0) | 2 (2) — skin tape stripping sites
skin dryness (General disorders) | 0 (0) | 3 (3) | 0 (0)
skin itching (General disorders) | 0 (0) | 6 (6) | 4 (4)
skin burning sensation (General disorders) | 0 (0) | 1 (1) | 1 (1)
skin tingly sensation (General disorders) | 0 (0) | 2 (2) | 0 (0)
skin peeling (General disorders) | 0 (0) | 1 (1) | 0 (0)
urticaria (General disorders) | 0 (0) | 1 (2) | 0 (0)
upset stomach/indigestion (General disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (General disorders) | 0 (0) | 1 (1) | 0 (0)
hematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) — post blood draws
skin erythema (redness) (General disorders) | 5 (5) | 10 (10) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03145259/Prot_SAP_000.pdf